CLINICAL TRIAL: NCT01039311
Title: Optical Coherence Tomography: An Adjunct to Flexible Bronchoscopy in the Diagnosis of Lung Cancer
Acronym: OCT
Status: Terminated | Type: Observational
Why Stopped: Unable to enroll subjects
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 14370
Record Dates: First submitted 2009-12-11; First posted 2009-12-24 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: Lung; cancer; bronchoscopy; optical; coherence; tomography
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Optical Coherence Tomography: Examine OCT images and compare them to conventional biopsies in same subject.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Obtain OCT images.
  Other Names: Imalux Niris

SUMMARY:
Optical coherence tomography will be a feasible adjunct to flexible bronchoscopy, and provide images with good sensitivity and specificity to determine the presence of endobronchial malignancies.

DETAILED DESCRIPTION:
OCT could become a powerful tool in diagnostic pulmonary medicine, not only in the early recognition of lung cancer, but also in the evaluation and monitoring of microstructures in the lower respiratory tract that are affected by other inflammatory or invasive disease processes. Initially, OCT could be used to guide the location of biopsies which would likely provide increased specificity to traditional bronchoscopy. However, if the sensitivity and specificity of OCT images are comparable to histologic specimens, this technology may in the future provide a non-invasive "optical biopsy", which could potentially obviate the need for conventional biopsies in patients with high risks for complications, such as bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-99 years of age
* Presence of an endobronchial mass
* Need for flexible bronchoscopy, with endobronchial biopsies

Exclusion Criteria:

* PCO2 > 47 mm Hg, and/or long term Oxygen therapy
* Unwillingness to undergo fiberoptic bronchoscopy
* Coagulopathy, defined as a platelets count < 100.000/mm3, or an INR> 1.4, or known clinical bleeding disorder
* Therapy with anticoagulant, including Coumadin and Clopidogrel
* Renal dysfunction, defined as a Creatinine > 2 mg/dl
* Life-threatening arrhythmias, or history of myocardial infarction within 6 months
* Cerebrovascular Accident within the preceding 6 months
* Facial abnormality preventing safe introduction of the bronchoscope
* Uncontrolled hypertension
* Active liver disease
* Pregnancy or Breastfeeding
* Prisoners
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 18-99 with the presence of of an endobronchial mass.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
OCT image sensitivity and specificity in diagnosis of lung cancer. | Every 3 months

SECONDARY OUTCOMES:
Feasibility and safety of obtaining OCT images during flexible bronchoscopy. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Keddissi, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Michel RG, Kinasewitz GT, Fung KM, Keddissi JI. Optical coherence tomography as an adjunct to flexible bronchoscopy in the diagnosis of lung cancer: a pilot study. Chest. 2010 Oct;138(4):984-8. doi: 10.1378/chest.10-0753. Epub 2010 May 14. PMID 20472863